CLINICAL TRIAL: NCT05278260
Title: Hydrogen Rich Water to Mitigate Acute Mucositis During Radiation Therapy
Brief Title: Hydrogen-rich Water and Treatment of Mucositis Caused by Radiation Therapy in Head and Neck Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: DrinkHRW (Unknown)
Responsible Party: Principal Investigator, Clare Moran, Survivorship Program Coordinator - Department of Radiation Oncology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SBU-HYDROGEN-HN-RT
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Mucositis Oral
Keywords: head and neck cancer; radiation therapy; supportive care
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms | interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control
- Active (Experimental)
  Interventions: Dietary Supplement: Hydrogen tablets

INTERVENTIONS:
Dietary Supplement: Hydrogen tablets — Participants will drink up to 1000 ml (34 fl. oz.) of water daily supplemented with a tablet that releases molecular hydrogen, for the duration of the radiation therapy
  Arms: Active
Dietary Supplement: Control — Participants will drink up to 1000 ml (34 fl. oz.) of water daily supplemented with a tablet that does not release any molecular hydrogen, for the duration of the radiation therapy
  Arms: Control

SUMMARY:
This study explores the effects of hydrogen-rich water on alleviating the radiation-induced acute mucositis in head and neck cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a biopsy proven head and neck cancer, early or advanced stage, primary or recurrent tumor,
* Planning to receive daily fractionated radiotherapy for over 4 weeks' duration
* Karnofsky Performance Score (KPS) of at least 70
* Able to describe pain
* Able to swallow food and water
* Able to sign consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop grade 3 oropharyngeal mucositis | 3 months after completing radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Mani, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No